CLINICAL TRIAL: NCT03576911
Title: Coenzyme Q10 in the Amelioration of Cognitive Deficits and Symptoms in Schizophrenia and Schizoaffective Disorder
Brief Title: A Randomised Controlled Trial of Coenzyme Q10 in Patients With Schizophrenia and Schizoaffective Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Liverpool John Moores University (Other); Royal Liverpool University Hospital (Other Government)
Responsible Party: Principal Investigator, Michael Gill, MD, Professor, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRFSJ0087
Record Dates: First submitted 2018-06-21; First posted 2018-07-05 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coenzyme Q10 (Experimental): 100mg CoQ10 capsule taken orally three times per day for 6 months
  Interventions: Dietary Supplement: Coenzyme Q10
- Placebo (Placebo Comparator): Placebo capsule taken orally three times per day for 6 months
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10
  Other Names: Ubiquinone Q10; Ubidecarenone
  Arms: Coenzyme Q10
Other: Placebo
  Arms: Placebo

SUMMARY:
The study is a randomised placebo controlled trial of Coenzyme Q10 (CoQ10) vitamin supplementation in a sample of patients with schizophrenia or schizoaffective disorder. CoQ10 is produced in the mitochondria of our cells, and is involved in the production of energy. However, some people do not produce enough CoQ10, which can result in difficulties with concentration and memory, depressive symptoms, low energy levels and high blood pressure. The study will examine the impact of taking oral CoQ10 supplementation on patients with schizophrenia and schizoaffective disorder.

DETAILED DESCRIPTION:
Coenzyme-Q10 (CoQ10) is an essential cofactor in the mitochondrial electron-transport-chain in addition to being a potent lipophilic antioxidant. Deficits in CoQ10 status have been linked to cardiovascular disease, cognitive decline, fatigue, and depression. CoQ10 supplementation may have a potential therapeutic value for patients with schizophrenia and schizoaffective disorder. This is a double-blind, placebo-controlled, randomised trial that will compare neurocognitive performance and symptoms of schizophrenia and schizoaffective disorder in participants randomised to active CoQ10 compared to scores from participants who received placebo. CoQ10 will be administered at a dose of 300mg/day, delivered in 3 doses of 100mg each. Participants will take CoQ10/placebo for 6 months. At three time points (baseline, 3 months and 6 months) each participant completes a neurocognitive and psychological battery of assessments. Blood pressure is monitored, and blood samples to assess mitochondrial function and plasma CoQ10 status are taken at each assessment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia or schizoaffective disorder

Exclusion Criteria:

* Current substance abuse
* History of epilepsy/seizures
* Head injury with loss of consciousness (>3 minutes)
* Taking warfarin or blood thinning medication
* Uncontrolled thyroid dysfunction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline attention | 6 months post-supplementation initiation/Directly following study treatment period
  Change from baseline attention as measured by Continuous Performance Test, identical pairs version (CPT-IP)
Change from baseline working memory performance | 6 months post-supplementation initiation/Directly following study treatment period
  Change from baseline working memory performance as measured by Cambridge Neuropsychological Test Automated Battery (CANTAB) spatial working memory task.
Change from baseline working memory performance | 6 months post-supplementation initiation/Directly following study treatment period
  Change from baseline working memory performance as measured by Letter Number Sequencing of Wechsler Memory Scale-III.

SECONDARY OUTCOMES:
Change from baseline processing speed | 6 months post-supplementation initiation/Directly following study treatment period
  Change from baseline processing speed as measured by Verbal Fluency Task
Change from baseline processing speed | 6 months post-supplementation initiation/Directly following study treatment period
  Change from baseline processing speed as measured by Trail Making Task
Change from baseline energy levels | 6 months post-supplementation initiation/Directly following study treatment period
  Change from baseline energy levels as measured by Functional Assessment of Chronic Illness Therapy - fatigue scale. Higher scores on this scale (total score range: 0-52) indicate better outcome.
Change from baseline depression levels | 6 months post-supplementation initiation/Directly following study treatment period
  Change from baseline depression levels as measured by Beck's Depression Inventory II
Change from baseline anxiety levels | 6 months post-supplementation initiation/Directly following study treatment period
  Change from baseline anxiety levels as measured by Beck's Anxiety Inventory
Change from baseline negative symptoms of avolition, asociality, blunted affect and alogia levels | 6 months post-supplementation initiation/Directly following study treatment period
  Change from baseline negative symptoms of avolition, asociality, blunted affect and alogia levels as measured by Brief Negative Symptoms subscales
Change from baseline blood pressure (systolic and diastolic) | 6 months post-supplementation initiation/Directly following study treatment period
  Change from baseline blood pressure (systolic and diastolic)
Change from baseline plasma CoQ10 levels | 6 months post-supplementation initiation/Directly following study treatment period
  Change from baseline plasma CoQ10 levels
Change from baseline mitochondrial function | 6 months post-supplementation initiation/Directly following study treatment period
  Change from baseline mitochondrial function as measured by plasma lactate levels

OTHER OUTCOMES:
Change from baseline self-reported quality of life | 6 months post-supplementation initiation
  Change baseline self-reported quality of life (WHOQOL-Bref)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gill, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- Clinical Research Facility, St James's Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maguire A, Mooney C, Flynn G, Ferguson Y, O'Keane V, O'Rourke D, McMonagle T, Heaton R, Phillips S, Hargreaves I, Gill M, Hargreaves A. No Effect of Coenzyme Q10 on Cognitive Function, Psychological Symptoms, and Health-related Outcomes in Schizophrenia and Schizoaffective Disorder: Results of a Randomized, Placebo-Controlled Trial. J Clin Psychopharmacol. 2021 Jan/Feb 01;41(1):53-57. doi: 10.1097/JCP.0000000000001330. PMID 33347024